CLINICAL TRIAL: NCT04488276
Title: Perceived Effects of Second-hand Smoke on a Pregnant Woman: A Phenomenological Study
Brief Title: Effects of Second-hand Smoke on a Pregnant Woman
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Maternal, Neonatal and Child Health Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: AC19107
Record Dates: First submitted 2020-04-17; First posted 2020-07-27 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Post Partum; Pregnancy Related
Keywords: Second hand smoke; Smoking fathers; Pregnant women; Post partum women

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: Non smoking pregnant and post-partum women
  Interventions: Other: In-depth interviews
- Smoking fathers: Expectant or new fathers who smoke
  Interventions: Other: In-depth interviews

INTERVENTIONS:
Other: In-depth interviews — In-depth interviews will be conducted to understand how smoking partners of pregnant women perceive risks and behaviors related to SHS exposure and how can it be altered to decrease exposure of pregnant women to SHS. These will be conducted in peri-urban slums and rural settings of Rawalpindi district with expectant or new father who smoke and pregnant or new mothers exposed to SHS. Interview guide will be developed deductively as a result of the systematic review and will be piloted before its actual use. Trained interviewer will conduct in-depth interview using semi-structured interview guide and will record it with consent from respondents. This data will be transcribed and translated and coded by team of two researchers.

SUMMARY:
More than 40% of all pregnant women in Pakistan are exposed to second-hand smoke - causing approximately 17,000 still births in a year. In Pakistan only 1% of still births are attributed to women actively smoking during pregnancy, but for second-hand smoke the figure is 7%, largely due to the high numbers of pregnant women exposed to tobacco smoke in the home. Negative effects of Second-hand smoking (SHS) on maternal and fetal health are well established. In low and middle-income countries (LMICs) smoking inside the house is largely unrestricted adversely affecting pregnant women by exposure to SHS. SHS exposure in non-smoking pregnant women has increased the risk of stillbirth and congenital malformation along with behavioural and cognitive issues in children. Partner's support during pregnancy is important for developing a better maternal health. Therefore, a phenomenological research approach is appropriate for describing the essence of experience in terms of affective and emotional aspects. Phenomenology is an approach of creating phenomenological knowledge in a situation by describing implicit meaning of experience. The investigators therefore propose an epistemological approach of phenomenology.

DETAILED DESCRIPTION:
INTRODUCTION:

Different forms of tobacco such as cigarettes, water pipe, chewing paan, gutka and naswar are used in Pakistan. According to Global Adult Tobacco Survey (2014), overall prevalence of tobacco use in Pakistan is 19.1% (23.9 million adults). 7 out of 10 adults and 5 out of 10 children are exposed to second hand smoke in indoor workplace and at home. Second hand smoke (SHS) is strongly associated with exposure of non-smoking pregnant women to various toxicants which can harm the fetus and post partum harm infants and children. Effects of second-hand smoking during pregnancy include low birth weight, sudden infant death, acute and chronic respiratory symptoms, asthma and ear infection . In South and Southeast Asia, women have a higher rate of exposure to SHS than men whereby they are exposed in different places disproportionality, such as public transportation (62%), restaurants (56%) and at workplace (37%). In LMICs, smoking inside the home is unrestricted and pregnant women are adversely affected by exposure to SHS which increases the risk of stillbirth and congenital malformation. It is, therefore, important to avert negative consequences of pregnancies that are exposed to second-hand smoke.

BACKGROUND:

Previously researchers have tried to explore societal and cultural aspects of indoor smoking and exposure to SHS and attributed gender inequality and gendered power dynamics to women's failure to negotiate smoke-free homes. Additionally, several interventions have been found to be effective in changing smoking-related behavior, however, most do not provide think description of interventions to ascertain their theoretical basis. Therefore, examining the phenomenon of second-hand smoke with an in-depth understanding of social and cultural factors may help in describing smoking- and anti-smoking related behavior through qualitative exploration. Findings of this pioneering qualitative work can be utilized for designing an effective reduction strategy for tobacco use which can act as a conceptual framework for behavior change to reduce or eliminate the effects of second-hand smoke on pregnant women.

More than 40% of all pregnant women in Pakistan are exposed to second-hand smoke - causing approximately 17,000 still births in a year. In Pakistan only 1% of still births are attributed to women actively smoking during pregnancy, but for second-hand smoke the figure is 7%, largely due to the high numbers of pregnant women exposed to tobacco smoke in the home. Negative effects of Second-hand smoking (SHS) on maternal and fetal health are well established. In LMICs smoking inside the house is largely unrestricted adversely affecting pregnant women by exposure to SHS. SHS exposure in non-smoking pregnant women has increased the risk of stillbirth and congenital malformation along with behavioral and cognitive issues in children. Partner's support during pregnancy is important for developing a better maternal health. Therefore, a phenomenological research approach is appropriate for describing the essence of experience in terms of affective and emotional aspects. Phenomenology is an approach of creating phenomenological knowledge in a situation by describing implicit meaning of experience. The investigators therefore propose an epistemological approach of phenomenology.

Informed by the findings of the systematic review on the risk perception of second-hand smoke, an interview guide will be developed. Int depth interviews with expectant or new fathers who smoke (n=25-30) and their pregnant or post-partum partners exposed to SHS(n=10-15) will be conducted. Thematic analysis will then be done. In addition to presenting findings of research in traditional manner (themes), they will also be presented in more applied or ready-to-be-picked manner. It means that based on the findings of this study an evidence-informed conceptual framework will be developed to propose a behavior change communication intervention, which will target poor or risky behaviors to promote behavior modification that may result in positive maternal and fetal health outcomes.

This will be a qualitative study incorporating an initial stage of systematic review followed by a stage of in depth interviewing that will lead to development of the conceptual framework.

METHODOLOGY:

Stage I:

Search Strategy:

Firstly, a review protocol will be developed(followed by its registration in (PROSPERO) incorporating key terms and alternate search terms which are given below:

* Second hand smoke: Indirect smoke, involuntary smoke, passive smoke
* Perception: Opinion, Perspective, Experience
* Pregnancy: Pregnant woman, post-partum woman

These search terms will be used in different combinations to form search string with use of Boolean operators (AND, OR) and truncations. PubMed, Embase, Global Health and CINAHL will be searched systematically to identify and retrieve relevant data. Inclusion criteria are given below:

* Qualitative studies or mixed method studies
* Studies covering perception of effects of SHS on pregnancy

Database Search:

Two independent reviewers will implement the search strategy and compile extracted data in Microsoft Excel sheet. The PRISMA workflow will be employed to complete the search.

Quality Assessment:

Critical Appraisal Skills Programme (CASP) or Joanna Briggs Institute (JBI) tool will be used to critically appraise the research studies. Two reviewers will appraise and report the result independently.

Data Extraction:

Data will be extracted at two levels: first order construct (participant's quote) and second order constructs (researcher's interpretation).

Data Synthesis and Reporting:

Extracted data will be assembled into collective findings which will explain the phenomenon under study. The necessary information extracted from each included paper will be descriptive (regarding the participants, study type and characteristics, location, setting, year, main topic, etc.), methods, type of analysis, findings, and original quotations. Thematic analysis of data will be employed. Double data extraction, which is considered the golden standard, will be employed. As a first step initial codes according to the analytical approach will be created. As the analysis progresses, it might be that some findings form a code, or they might become a code combined with other findings. It might also require for some codes to be collapsed in order to form another code or (sub)theme. The data, once compiled and analyzed, will also be available for depositing and publishing on an open research data platform.

Stage 2:

Settings:

Study will be conducted in Urban and peri-urban settings of Rawalpindi district.

Research Design:

Our qualitative approach will include in depth interviewing.

Sampling:

Purposive sampling will be employed to select potential respondents from different socio-economic and education background. Though number of respondents will be determined by theoretical saturation, but for planning purpose the investigators will recruit 25-30 smokers and 10-15 non-smoking pregnant or post-partum women.

Potential Respondents:

Community gatekeepers and lady health workers will be used to identify expectant and new fathers, who are active smokers, along with pregnant and post-partum women who are exposed to SHS.

Data Collection:

Interview guide will be developed deductively as a result of the systematic review and will be piloted before its actual use. Guide will be revised based on the experience of pilot interview or as data collection proceeds. Trained interviewer will conduct in-depth interview using semi-structured interview guide and will record it with consent from respondents. Later, services of professional transcriber and translator will be taken and data will be coded by team of two researchers.

Data Analysis:

Inductive approach of extracting codes from the textual data will be utilized. Initial coding structure will be developed and discussed and same will undergo several iterations based on the review of other transcripts. Final coding scheme will be uniformly applied to all interview transcripts. Inductive thematic analysis approach will be used to identify behaviors and methods of behavior development. Narrative account on lived experiences will help us to contextualize key behavior within cultural and social context of the Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Non smoking pregnant women exposed to second hand smoke
* Non smoking women in post partum period exposed to second hand smoke
* Expectant or new fathers who smoke
* Respondents residing in rural and per urban slums of Rawalpindi district
* Respondents who consent to participate in the study

Exclusion Criteria:

* Non smoking fathers
* Women not exposed to second hand smoke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Number of Participants:
  Sample size will be based on the point of theoretical saturation, although at least 25-30 interviews will be conducted with fathers who are smokers and 10-15 with non-smoking pregnant or post-partum women exposed to second hand smoke.
  - Identifying participants: Community gatekeepers and lady health workers will be used to identify expectant and new fathers, who are active smokers, along with pregnant and post-partum women who are exposed to SHS.
  - Consenting participants A written and signed consent form will be obtained from all of the participants.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of pregnant women exposed to SHS | six months
  In depth interviews will be conducted using a semi structured interview guide
proportion of smoker husbands with adequate knowledge of effects of SHS on pregnancy | six months
  In depth interviews will be conducted with assess the knowledge using a semi structrured interview guide

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tabish Hazir, MBBS, FRCPCH, Principal Investigator — Maternal, Neonatal and Child Health Research Network
Locations (1):
- MNCHRN, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided